CLINICAL TRIAL: NCT04003064
Title: Heavy Metals' Influence on Early Pregnancy Through Oxidative Stress
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HML2019
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-05

CONDITIONS: Spontaneous Abortion; Oxidative Stress
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — blood and urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood — 3ml blood

SUMMARY:
Patients with diagnosis of spontaneous abortion are enrolled in the cohort, in the cohort of patients who met the criteria, 3ml of whole blood intravenous and 5ml of urine were taken for heavy metal level examnation. Part of the villi tissue was sent for genetic testing, and the results were traced. In addition, about 10g of villi tissue was frozen for testing. Patients with normal genetic results of villi tissue will have villus samples go through oxidative stress level detection.

DETAILED DESCRIPTION:
From May 1, 2019, patients with diagnosis of spontaneous abortion are enrolled in the cohort, exclusion criteria were: not long-term residents in Peking; Inconvenient for following up; Long-term of drug use; Cesarean section scar pregnancy and other high-risk pregnancy; Diagnosis of pregnancy beyond 12 weeks.

In the cohort of patients who met the criteria, 3ml of whole blood intravenous and 5ml of urine were taken on the day of admission for curettage and suction, and the levels of heavy metals were tested. Part of the villi tissue was sent for genetic testing, and the results were traced. In addition, about 10g of villi tissue was frozen for testing. Patients with normal genetic results of villi tissue will have villus samples go through oxidative stress level detection.

ELIGIBILITY:
Inclusion Criteria:

1) the length of fetal bud is equal to or greater than 7 mm and there is no cardiac activity; 2) the maximum zh diameter of the pregnancy sac is equal to or greater than 25mm, and there is no fetal heart beat; 3) an embryo with no heartbeat at 2 weeks or more after ultrasound examination showing a pregnancy sac without yolk sac; 4) embryos without heartbeat for 11 days or longer after ultrasonography showed the yolk sac as a type pregnancy sac.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Exclusion Criteria:
  not long-term residents in Peking; Inconvenient for following up; Long-term of drug use; Cesarean section scar pregnancy and other high-risk pregnancy; Diagnosis of pregnancy beyond 12 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
oxident stress level | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xinyan U Liu, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No